CLINICAL TRIAL: NCT06807762
Title: Phase I Clinical Trial to Assess Tolerability, Safety, and Pharmacokinetics of Extrato de Cannabis Sativa GreenCare 79.14 mg/mL - Drops Solution - in Healthy Research Participants of Both Sexes in a Fed State
Brief Title: Safety and Pharmacokinetics of Extrato de Cannabis Sativa GreenCare
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GreenCare Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GreenCare-ExtratoCannabis-0124; 131.001.23 (Other: Synvia Clinical | CAEP)
Record Dates: First submitted 2025-01-17; First posted 2025-02-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extrato de Cannabis sativa GreenCare 79.14 mg/mL (Experimental): Concentration unit: 79.14 mg/mL
  Interventions: Drug: Cannabis oil

INTERVENTIONS:
Drug: Cannabis oil — Healthy subjects will be treated with a solution of Cannabis sativa extract diluted in MCT oil, at doses ranging from 39.62 mg to 791.4 mg. This protocol will be divided into two stages:
  Stage 1 - Determination of the Maximum Tolerated Dose (MTD): Participants (n=60) will be dynamically randomized and will receive Cannabis sativa extract (GreenCare, 79.14 mg/mL) as a single dose after breakfast, with doses ranging from 39.62 mg to 791.4 mg.
  Stage 2 - Assessment of the MTD: All participants (n=12) will receive the MTD determined in Stage 1, administered in two daily doses for 14 consecutive days.
  Other Names: Extrato de Cannabis sativa GreenCare 79.14 mg/mL

SUMMARY:
The goal of this Phase I clinical trial is to assess the pharmacokinetic availability and safety and tolerability profile of Extrato de Cannabis sativa GreenCare 79.14 mg/mL. The main question it aims to answer is:

• Is the Extrato de Cannabis sativa GreenCare 79,14 mg/mL safe?

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years, inclusive;
* Body weight ≥ 50 kg and BMI between 18.5 and 30 kg/m2, inclusive;
* Be healthy according to medical history, i.e., have laboratory test results within normal ranges and/or any deviations from normal classified as clinically insignificant;
* Be exclusively participating in this clinical study during the research period;
* Understand and comply with the protocol requirements and consent to participate in the study by signing the Informed Consent Form (ICF) approved by an Ethics Committee (EC).

Exclusion Criteria:

Having participated in any experimental study or ingested any experimental drug within 1 (one) year prior to the start of this study;

* Inability to use oral medication and/or cooperate with investigators due to cognitive impairment or mental state;
* Reported allergy to any component of Cannabis sativa extract 79.14 mg/mL;
* Personal or first-degree family history of schizophrenia, bipolar affective disorder, psychotic symptoms, suicidal ideation, planning and/or attempt, and/or severe uncontrolled psychiatric comorbidities, at the discretion of the principal investigator;
* Donated blood within four (4) months prior to signing the Informed Consent Form (ICF);
* Being pregnant, breastfeeding, intending to become pregnant during the study period, or having a positive result for urinary β-HCG testing;
* Reported use of Cannabis and/or its derivatives for any purpose in the past 6 months;
* Personal history of Cannabis use disorder and/or other illicit drug use disorder;
* Personal history of alcohol, tobacco, opioid, benzodiazepine, barbiturate, and/or other substance use disorders, such as St. John's Wort;
* Smokers or ex-smokers who quit less than 6 months ago;
* Consumed alcoholic beverages within 24 hours before the study confinement period;
* Any condition that prevents participation at the discretion of the investigator;
* Dietary habits that prevent ingestion of the diet provided during the study;
* Any clinical or laboratory finding or therapy that, at the investigator's discretion, may place the participant at risk or interfere with study objectives or outcomes;
* Non-compliance with the complete ingestion of the diet provided - determination at the discretion of the responsible physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the Maximum Tolerated Dose (MTD) of Cannabis sativa Extract GreenCare 79,14 mg/mL | Up to 5 days

SECONDARY OUTCOMES:
Frequency, intensity, and severity of adverse events | Up to 5 days
Plasma concentrations of CBD and THC | Up to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Pacheco, MD, Principal Investigator — Synvia Clinical | CAEP
Locations (1):
- GreenCare Pharma, Vinhedo, São Paulo, Brazil